CLINICAL TRIAL: NCT05433272
Title: A Randomized, Double-Blind, Active-controlled Phase Ⅲ Clinical Trial to Evaluate the Immunogenicity and Safety of One Booster Dose of Trivalent COVID-19 Vaccine (Vero Cell), Inactivated in Healthy People in Colombia
Brief Title: Immunogenicity and Safety Study of One Booster Dose of Trivalent COVID-19 Vaccine (Vero Cell), Inactivated
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinovac Biotech (Colombia) S.A.S. (Industry)
Collaborators: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-tnCOV-3003
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Trial group of participants have received two doses of CoronaVac® (Experimental): 400 participants have received two doses of CoronaVac® at least 3 months prior to this study ,including 150 participants aged 3-17 years old,125 participants aged 18-59 years old and 125 participants aged 60 years and above,will receive one booster dose of trivalent COVID-19 vaccine.
  Interventions: Biological: Trivalent COVID-19 Vaccine (Vero Cell), Inactivated, Prototype Strain, Delta Strain and Omicron Strain
- Control group of participants have received two doses of CoronaVac® (Active Comparator): 400 participants have received two doses of CoronaVac® at least 3 months prior to this study ,including 150 participants aged 3-17 years old,125 participants aged 18-59 years old and 125 participants aged 60 years and above,will receive one booster dose of CoronaVac®.
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- Trial group of participants have received three doses of CoronaVac® (Experimental): 300 participants have received three doses of CoronaVac® at least 3 months prior to this study ,including 150 participants aged 18-59 years old and 150 participants aged 60 years and above,will receive one booster dose of trivalent COVID-19 vaccine.
  Interventions: Biological: Trivalent COVID-19 Vaccine (Vero Cell), Inactivated, Prototype Strain, Delta Strain and Omicron Strain
- Control group of participants have received three doses of CoronaVac® (Active Comparator): 300 participants have received three doses of CoronaVac® at least 3 months prior to this study ,including 150 participants aged 18-59 years old and 150 participants aged 60 years and above,will receive one booster dose of CoronaVac®.
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: Trivalent COVID-19 Vaccine (Vero Cell), Inactivated, Prototype Strain, Delta Strain and Omicron Strain — The Trivalent COVID-19 Vaccine (Vero Cell), Inactivated, Prototype Strain, Delta Strain and Omicron Strain was developed by Sinovac Life Science Ltd. The antigen content of trivalent COVID-19 vaccine is a total of 18μg/0.5 ml, including 1200 SU/6 µg/0.5 ml for Prototype strain, 1200 SDU/6 µg/0.5 ml for Delta strain, and 1200 SOU/6 µg/0.5 ml for Omicron strain. The routine of administration is Intramuscular injection into deltoid region.
  Other Names: Trivalent COVID-19 vaccine
  Arms: Trial group of participants have received three doses of CoronaVac®; Trial group of participants have received two doses of CoronaVac®
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — The COVID-19 Vaccine (Vero Cell),Inactivated was manufactured by Sinovac Life Science Ltd.The antigen content of the active-controlled vaccine (CoronaVac) is 600 SU/3 µg/0.5 ml.The routine of administration is Intramuscular injection into deltoid region.
  Other Names: CoronaVac®
  Arms: Control group of participants have received three doses of CoronaVac®; Control group of participants have received two doses of CoronaVac®

SUMMARY:
This is a randomized, double-blind, active-controlled phase Ⅲ clinical trial.The purpose of this study is to evaluate the immunogenicity and safety of one booster dose of trivalent COVID-19 vaccine (vero cell), inactivated, prototype strain, delta strain and omicron strain in healthy people aged 3 years old and above and have completed two or three doses of CoronaVac® in Colombia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, and active-controlled Phase Ⅲ bridging clinical trial of 1,400 subjects aged 3 years and above and have completed two or three doses of CoronaVac at least 3 months prior to this study.After enrollment, subjects will be randomly assigned into 2 groups at a ratio of 1:1 to receive one dose of trivalent COVID-19 vaccine or CoronaVac®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people aged 3 years and above who have completed two or three doses of CoronaVac at least 3 months (≥ 90 days) before (3-8 weeks interval for the first and second dose of CoronaVac, and ≥3 months interval for the second and third dose);
* Participants (and/or their legal guardians for pediatric population) are able to understand and sign the informed consent voluntarily;
* Pregnancy and contraception:

Female participants of childbearing potential (post-menarche and pre-menopause that has not been undergone any sterilization surgery), who have a negative pregnancy test on the day of booster vaccination in the present study, has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the day of vaccination, and agree to continue adequate contraception through 3 months following the booster vaccination and are not currently breastfeeding; Male participants of childbearing potential who agree to use adequate contraception through 3 months following the booster vaccination (and/or your female partner agree to use an acceptable method of birth control), which include refrain from donating sperm;

Note 1 :Adequate contraception is defined as consistent and correct use of an approved contraceptive method in accordance with the product label. For example:

* Barrier method (such as condoms, diaphragm, or cervical cap) used in conjunction with spermicide
* Intrauterine device
* Prescription hormonal contraceptive taken or administered via oral (pill), transdermal (patch), subdermal, or IM route
* Sterilization of a female participant's monogamous male partner prior to entry into the study Note 2 : Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

  * Participants are able to comply with study procedures based on the assessment of the Investigator;
  * Participants willing to provide verifiable identification (following the local regulations), to be contacted, and to contact the investigator during the study period.

Exclusion Criteria:

* History of confirmed infection of SARS-CoV-2 within 3 months prior to study vaccination；
* With positive test result of SARS-CoV-2 antigen during screening visit;
* Any prior administration of another investigational COVID-19 vaccine or other licensed COVID-19 vaccines, or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Known allergy to vaccines or vaccine ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Serious chronic disease, including but not limited to serious cardiovascular disease, hypertension and diabetes that drugs cannot control, hepatorenal disease, malignant tumor, etc;
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* Significant chronic central nervous system diseases or neuromuscular disorders, psychosis or severe cognitive behavioral disorder, in the opinion of the investigator, including but not limited to epilepsy, autism spectrum disorder, intellectual disabilities;
* History of autoimmune and/or hematological diseases (including but not limited to systemic lupus erythematosus, thyroidectomy, autoimmune thyroid disease, hematological malignancy, asplenia, functional asplenia, or splenectomy resulting from any condition);
* History of bleeding disorders (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture;
* Receipt of blood/plasma products or immunoglobulins in the past 3 months before vaccination in this study;
* Participation in other studies involving study intervention within 30 days prior to vaccination in this study;
* Receipt of attenuated live vaccines in the past 14 days prior to vaccination in this study;
* Receipt of inactivated or subunit vaccines in the past 7 days prior to vaccination in this study;
* Emerging of chronic diseases or acute exacerbation of stable chronic diseases (including but not limited to asthma, migraine, gastrointestinal disorder, etc.) within 30 days prior to vaccination in this study;
* Acute febrile illness, or body temperature ≥37.8°C on the day of vaccination; enrollment could be considered if the fever is absent for 72 hours prior to vaccination;
* According to the investigator's judgment, the participant has any other factors that might interfere with the clinical trial results or pose additional risk to the participant due to participation in the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain | At 14 days after one booster dose
  Geometric Mean Titer (GMT) of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac
Seroconversion rate of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain | At 14 days after one booster dose
  Seroconversion rate of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac
GMT of the neutralizing antibody to SARS-CoV-2 Prototype strain | At 14 days after one booster dose
  GMT of the neutralizing antibody to SARS-CoV-2 Prototype strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac.
Seroconversion rate of the neutralizing antibody to SARS-CoV-2 Prototype strain | At 14 days after one booster dose
  Seroconversion rate of the neutralizing antibody to SARS-CoV-2 Prototype strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac.

SECONDARY OUTCOMES:
Seropositive rate of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain | At 14 days after one booster dose
  Seropositive rate of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac.
Geometric Mean Fold Rise (GMFR) of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain | At 14 days after one booster dose
  Geometric Mean Fold Rise (GMFR) of the neutralizing antibody to SARS-CoV-2 Delta strain and Omicron strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac
Seropositive rate of the neutralizing antibody to SARS-CoV-2 Prototype strain | At 14 days after one booster dose
  Seropositive rate of the neutralizing antibody to SARS-CoV-2 Prototype strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac
GMFR of the neutralizing antibody to SARS-CoV-2 Prototype strain | At 14 days after one booster dose
  GMFR of the neutralizing antibody to SARS-CoV-2 Prototype strain at 14 days after one booster dose of trivalent COVID-19 vaccine or CoronaVac.
Occurrence, intensity, duration, and relationship of solicited local and systemic Adverse Reactions (ARs) | Within 7 days after booster vaccination
  Occurrence, intensity, duration, and relationship of solicited local and systemic Adverse Reactions (ARs) within 7 days after booster vaccination.
Occurrence, intensity, duration, and relationship of unsolicited ARs | within 28 days after booster vaccination
  Occurrence, intensity, duration, and relationship of unsolicited ARs within 28 days after booster vaccination.
Occurrence and relationship of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | Within 6 months after booster vaccination
  Occurrence and relationship of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) within 6 months after booster vaccination.

OTHER OUTCOMES:
Seropositive rate of neutralizing antibody | At 3 and 6 months after the booster dose
  Seropositive rate of neutralizing antibody to SARS-CoV-2 Prototype strain, Delta strain and Omicron strain at 3 and 6 months after the booster dose of trivalent COVID-19 vaccine or CoronaVac.
GMT of neutralizing antibody | At 3 and 6 months after the booster dose
  GMT of neutralizing antibody to SARS-CoV-2 Prototype strain, Delta strain and Omicron strain at 3 and 6 months after the booster dose of trivalent COVID-19 vaccine or CoronaVac.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Cadena, Doctor, Principal Investigator — Clinica de la Costa
Locations (1):
- Clinica de la Costa, Barranquilla, Colombia